CLINICAL TRIAL: NCT05111873
Title: Effects of Multimodal Treatment of Headache in a Day Clinic Service: a Prospective Case-crossover Study
Brief Title: Effects of Multimodal Treatment of Headache in a Day Clinic Service
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Other Study IDs: BB004/21
Record Dates: First submitted 2021-07-12; First posted 2021-11-08 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: Headache Disorders
Keywords: multimodal treatment; quality of life; day clinic service
MeSH Terms: conditions — Headache Disorders | interventions — Combined Modality Therapy

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- waiting-list control: Participants enquired prior to the treatment appointment in the neurological day clinic service, no intervention
- post-treatment group: Participants enquired after the treatment in the Neurological day clinic service
  Interventions: Other: multimodal treatment

INTERVENTIONS:
Other: multimodal treatment — combination of medical consultations, psychological therapy, physiotherapy, occupational therapy, disease specific education und progressive muscle relaxation
  Groups: post-treatment group

SUMMARY:
The observational study aims to investigate the effects of a multimodal treatment program for headache patients in a day clinic service. The setting provides one week of treatment including a combination of medical consultation, physiotherapy, psychological therapy, occupational therapy, progressive muscle relaxation and disease specific education.

Outcome measures are the disease-specific impact on daily activities, general quality of life, psychological impact and headache frequency. Moreover, the study sought to identify parameters that best predict efficacy of the intervention. Therefore, standardized questionnaires are established in three points in time, to evaluate the pre- and post-treatment status.

DETAILED DESCRIPTION:
duration of treatment: 5 days; first questionnaire (V0): minimal 4 weeks prior to the treatment appointment; second questionnaire (V1): on the first day of the treatment program; third questionnaire (V2 / Follow up): 3 month (+- 6 weeks) after finishing the treatment; data collection through patient self-report; Follow-up via mail

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of a headache disorder
* written informed consent for collecting and analysing data and conducting a follow-up evaluation

Exclusion Criteria:

* premature interruption of the treatment
* repeated treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients seen in the neurological day clinic service will be screened for eligibility.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-02-15 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
Change of Veterans RAND 12 Item Health Survey (VR-12) mental health score | 4 weeks prior to treatment appointment, day 1 of treatment, 3 month after the treatment
  questionnaire, patient self-report, 12 questions, minimum value: 12 points, maximum value: 54 points, physical and mental health component summary score compared to a t-score with a mean value of 50 and standard deviation of 10

SECONDARY OUTCOMES:
Change of Depression Anxiety and Stress Scale (DASS) | 4 weeks prior to treatment appointment, day 1 of treatment, 3 month after the treatment
  questionnaire, patient self-report, 21 questions, 7 questions per subscale (Depression, Anxiety and Stress), minimum value: 0 points, maximum value: 21 points per subscale, higher score = worse outcome
Change of Headache Impact Test (HIT6) | 4 weeks prior to treatment appointment, day 1 of treatment, 3 month after the treatment
  questionnaire, patient self-report, minimum value: 36 points, maximum value: 78 points, higher score = worse outcome
Change of Pain intensity | 4 weeks prior to treatment appointment, day 1 of treatment, 3 month after the treatment
  average pain intensity in the last month, scale 1 to 10, higher score = worse outcome
Change of Headache frequency | 4 weeks prior to treatment appointment, day 1 of treatment, 3 month after the treatment
  in days per month, referring to the last month, minimum value: 0 days/month, maximum value: 30 days/month
Change of Veterans RAND 12 Item Health Survey (VR-12) physical health score | 4 weeks prior to treatment appointment, day 1 of treatment, 3 month after the treatment
  questionnaire, patient self-report, 12 questions, minimum value: 12 points, maximum value: 54 points, physical and mental health component summary score compared to a t-score with a mean value of 50 and standard deviation of 10

OTHER OUTCOMES:
Change of Veterans RAND 12 Item Health Survey (VR-12) single domains | 4 weeks prior to treatment appointment, day 1 of treatment, 3 month after the treatment
  questionnaire, patient self-report, 12 questions, minimum value: 12 points, maximum value: 54 points, physical and mental health component summary score compared to a t-score with a mean value of 50 and standard deviation of 10

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, Greifswald, Mecklenburg-Vorpommern, Germany